CLINICAL TRIAL: NCT04543448
Title: Investigation the Effect of Cervical Mobilization on Balance and Plantar Pressure Distribution in Multiple Sclerosis Patients: A Randomized Crossover Controlled Study
Brief Title: Effect of Cervical Mobilization on Balance and Plantar Pressure Distribution in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuba Maden, Principal Investigator, clinical research, Hasan Kalyoncu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/0107
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis; Muscle Spasticity; Pressure Area; Cervical Region Disorder Nos
Keywords: cervical region; multiple sclerosis; muscle spasticity; manual therapy; cervical spine; Plantar pressure
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Participants are grouped randomly. First group and second group are applied different rehabilitation programs. Both of group is rest four weeks. Than second group is applied first group's rehabilitation program and first group is applied second group's rehabilitation program.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Rehabilitation (Other): Traditional Rehabilitation program was included strengthening exercises for the muscles needed, balance and coordination exercises according to the individual's level, stretching for the lower limbs in all individuals. Indıvıduals participated in 2 training sessions per week for 4 weeks. Each training session consisted of a 5-minute non-balance coordination exercise, a 30-minute balance and coordination exercise, a 10-minute stretching and strengthing.
  Interventions: Other: Traditional Rehabilitation for multiple sclerosis
- Cervical Mobilization (Experimental): Cervical Mobilization program, cervical mobilization techniques were applied to the patients for 30 minutes in addition to the traditional program. Cervical mobilization includes suboccipital relaxing techniques, myofascial muscle relaxing techniques for Levator scapula, trapezius, scalenes muscles. These techniques were applied bilaterally.
  Interventions: Other: Cervical mobilization for multiple sclerosis

INTERVENTIONS:
Other: Traditional Rehabilitation for multiple sclerosis — Traditional rehabilitation program include strengthening exercises for the muscles needed, balance and coordination exercises according to the individual's level, stretching for the lower limbs.
  Other Names: traditional rehabilitation
  Arms: Traditional Rehabilitation
Other: Cervical mobilization for multiple sclerosis — Cervical mobilization program include myofascial relaxation techniques and mobilization to cervical spine in addition to traditional program.
  Other Names: traditional rehabilitation+ cervical mobilization
  Arms: Cervical Mobilization

SUMMARY:
MS patients were randomly divided into traditional therapy and traditional therapy + cervical mobilization groups. While muscle strengthening, stretching, balance and coordination exercises were given to the traditional group, cervical mobilization was applied in addition to these in cervical group. Patients received treatments twice a week for 4 weeks. The effect of the applied treatment on the tonus and plantar pressure distribution was analyzed. Treatments were interrupted for 4 weeks and the groups continued with the treatment they did not receive (crossover design). The group that received traditional treatment in the first period completed traditional + cervical mobilization, and the other group with traditional + cervical mobilization traditionally completed the treatment.

DETAILED DESCRIPTION:
Cervical region is rich in terms of muscle spindle and reseptors. When this region is touched by physiotherapists, muscle spindles is activited. The cervical region is parasympathetic area have common relaxed effect. Thus this part can be benefit to improvement of balance. As improve balance, the plantar pressure distribution of patients may change.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) score was between 2-5,
* According to the modified Ashworth Scale, spasticity is between 1 and 3,
* EDSS Cerebellar System Sub-Scale, Functional System Score ˃1,
* medical condition is stable and no medication changes were made in the last month,
* Vertebro-basillar test negative,
* Not have any other neurological disorder and orthopedic problem to prevent participation in this study
* A score of at least 24 from the Mini Mental Test,

Exclusion Criteria:

* presence of psychiatric or severe cognitive dysfunction,
* pregnancy,
* Having a neurological disease other than MS,

  * having had an attack in the last 3 months,
* Botulinum toxin application within the last 6 months,
* participating in physiotherapy program in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Change Plantar Pressure Distribution | Change from plantar pressure distribution at one month
  Pedobarography system was used for plantar pressure analyses. Pedobarography system contains screen, color printer, pressure sensor platform, remote control device, power unit, printer-to-platform and screen-to-platform connections. The maximum and mean pressure in the foot, the percentages of pressure values in the fore and rear of the foot, percentages of the total pressure falling to the foot were evaluated. As higher values mean higher load.
Change Balance | Change from plantar pressure distribution at one month
  Romberg test (RT) was performed on the patients with eyes closed and feet together. When the participant held it in one place, the test was terminated, oscillations began, or was likely to fall. Romberg test's maximum duration was 120 sec. RT is clinically used for vestibular problems.
  Sharpened Romberg (SR) was performed on a straight line with one leg behind the other leg, eyes open, leaving the arms sagging and without impairing the balance. Duration stop criteria were defined as the time that took a participant to dislocate the foot, reach the maximal duration of 30 sec, and contact the observer to avoid falling.
  Individuals' dynamic balance was evaluated with the Functional Reach Test (FRT). Individuals had requested their hands at 90 degrees by keeping the dominant arms' elbow straight on the wall. The test was performed as reaching forward without taking a step and losing the balance on the wall. The metacarpal bone level was marked in the start position and final position

SECONDARY OUTCOMES:
Change Modified ashworth scale | Change from Modified ashworth scale at one month
  Modified Ashworth Scale measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. The minimum value is 1 and the maximum value is 4. Whether higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: KEZBAN BAYRAMLAR, Prof. Dr., Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)